CLINICAL TRIAL: NCT04107896
Title: Efficacy of Silodosin in the Treatment of Symptomatic Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Maidul Islam, Resident,BSMMU, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No BSMMU/2017/9066
Record Dates: First submitted 2019-09-04; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silodosin (Experimental): 8 mg daily by mouth, 12 weeks
  Interventions: Drug: Silodosin
- Tamsulosin (Active Comparator): 0.4 mg daily by mouth, 12 weeks
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Silodosin — Cap silodosin
  Other Names: Rapasin
  Arms: Silodosin
Drug: Tamsulosin — Cap tamsulosin
  Other Names: Uromax
  Arms: Tamsulosin

SUMMARY:
In this study the investigators had evaluated the effectiveness SILODOSIN (8 mg daily orally) in Benign prostatic Hyperplasia in comparison to Tamsulosin (0.4 mg daily orally) in a randomized controlled trial design. Study population would be patients attending Urology OPD of BSMMU Hospital, Dhaka. Target sample size will be 136 evaluable patients in each group (assuming dropout rate 20%), suffering from Benign prostatic Hyperplasia .Subjects would be observed for 1 week without any drug. At the end of 1 week, they would be randomly allocated to Silodosin or Tamsulosin and treatment continued for 12 weeks. Interim follow-up visits would be at 1,4 and 12 weeks. USG confirmation of BPH would be required for recruitment. Effectiveness of the drugs would be assessed by International Prostate Symptom score, a quality of life (QoL) assessment done by a 7-point scale. Prostate weight/volume determination by USG, Change in post voidal residual urine (PVR) by USG and Changes in peak urine flow rate by uroflowmetry. Safety would be assessed by following up vital signs, treatment emergent adverse events and routine laboratory tests for drug safety.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is the most common cause of lower urinary tract symptoms in elderly men. Selective α1-adrenergic antagonists are now ﬁrst-line drugs in the medical management of BPH. This Hospital based randomized controlled clinical study designed to evaluate the efficacy of the new α1-blocker silodosin in the treatment of symptomatic benign prostatic hyperplasia (BPH).Ambulatory patients of age between 50 to 70 years, who were diagnosed as benign prostatic hyperplasia, were divided into two groups after fulfilling selection criteria. After informed consent & random sampling by lottery, silodosin 8 mg was given to group A (study) & tamsulosin 0.4 mg was given to group B (control). Total 149 patients were enrolled in this study but 8 patients were lost during follow up. Hence 141 patients completed the study, during the period of June 2017 to August 2018.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male patients between 50 to 70 years and had diagnosis of lower urinary tract symptoms associated with benign prostatic hyperplasia (BPH)
* International prostate symptoms score (IPSS)≥ 8
* Peak urinary flow rate (Qmax)<15ml/sec for a voided volume of 150 ml or more
* Post voidal residual urine volume ≥ 50 ml (by transabdominal ultrasonogram)
* Volume of prostate determine by transabdominal ultrasonogram ≥ 30 gm

Exclusion Criteria:

* History of prostate cancer/raised PSA>4 ng/ml
* Previous prostate surgery /Periurethral surgery.
* Patient undergone surgery to the bladder neck/Bladder neck contracture.
* Urethral stricture
* History of LUTS not due to benign prostatic hyperplasia (BPH).
* Postvoid residual urine volume of >150ml
* Bladder stone
* Active urinary tract infection which might affect micturition
* Large intravesical protrusion > 2 cm
* Known hypersensitivity or history of active substance abuse

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 141 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in IPSS & Quality of life (QoL) score | Screening visit, baseline visit, follow up visit at 1th, 4th and 12th week
  Effectiveness of silodosin in benign prostatic hyperplasia assessed by symptom relief as assessed by IPSS. The total score was taken as the sum of the seven individual symptom scores. Each individual scored 0-5 (0 = Minimum; 5 = Maximum as worse as can be), yielding a total between 0 and 35. The Storage sub score was taken as the sum of the three individual symptom scores (Range 0-15) & the Voiding sub score was taken as the sum of the four individual symptom scores (Range 0-20). Quality of life (QoL) score assessment was done on a 7-point scale 0-6 (0= Delighted; 6= Terrible).

SECONDARY OUTCOMES:
Changes in peak urine flow rate & post voidal residual urine (PVR) | Screening visit, baseline visit, follow up visit at 1th, 4th and 12th week
  Changes in peak urine flow rate by uroflowmetry & post voidal residual urine (PVR) by USG.

CONTACTS AND LOCATIONS:
Overall Officials: maidul islam, resident, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Maidul islam, Dhaka, Bangladesh